CLINICAL TRIAL: NCT06322940
Title: Effect of Dairy Product Matrices on Insulin Resistance in People with Overweight and Obesity and Prediabetes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Dairy Farmers of Canada (Other)
Responsible Party: Principal Investigator, Sergio Burgos, Associate Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2024-10463
Record Dates: First submitted 2024-02-29; First posted 2024-03-21 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: PreDiabetes; Overweight and Obesity
Keywords: Dairy products; Insulin sensitivity; Glucose metabolism; Insulin resistance
MeSH Terms: conditions — Prediabetic State; Overweight; Obesity; Insulin Resistance | interventions — Serving Size

STUDY DESIGN:
Intervention Model Description: Three treatment groups
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participant's study group will be coded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 2-3 servings of regular-fat milk (Experimental): Milk
  Interventions: Other: 250 mL serving size, 3.25% fat content
- 2-3 servings of regular-fat yogurt (Experimental): Yogurt
  Interventions: Other: 175 g serving size, ≥2% fat content
- 2-3 servings of regular-fat cheese (Experimental): Cheese
  Interventions: Other: 50 g serving size, ≥28% fat content

INTERVENTIONS:
Other: 250 mL serving size, 3.25% fat content — Milk
  Arms: 2-3 servings of regular-fat milk
Other: 175 g serving size, ≥2% fat content — Yogurt
  Arms: 2-3 servings of regular-fat yogurt
Other: 50 g serving size, ≥28% fat content — Cheese
  Arms: 2-3 servings of regular-fat cheese

SUMMARY:
The objective of the study is to determine the effect of dairy product matrices on insulin sensitivity in overweight and obese adults with prediabetes. Females and males (30-65 y) will be recruited from the greater Montreal area. Upon screening, those with prediabetes will complete a 2-wk run-in period in which participants will consume 1 serving/d of regular-fat dairy products (milk, yogurt, or cheese). Adherent participants will be randomized by sex into 1 of 3 groups: ≤1 serving/d of dairy (limited dairy) or 2-3 servings/d of reduced-fat or regular-fat dairy for 12 weeks. Participants will be instructed on how to incorporate foods into their diet to prevent changes in their body weight. The hyperinsulinemic-euglycemic clamp will be used before and after the intervention to document potential changes in insulin sensitivity as the primary outcome. In addition, glycemic variables, body composition, and cardiometabolic risk factors will be assessed as secondary outcomes. Adherence to intervention will be assessed at each visit by food diaries and a record of consumed dairy products.

DETAILED DESCRIPTION:
The randomized controlled trial will be preceded by a 2-week run-in period in which participants will consume 1 serving/day of regular-fat dairy. Following the run-in period, adherent participants will be randomly assigned to one of the three treatment groups (n=20 per group) in a 1:1:1 allocation ratio. Stratified permuted block randomization will ensure adequate balance among groups using a computer-generated list of random numbers. Due to the nature of the test products, participants cannot be blinded to the diet intervention. However, outcome assessors will be blinded to treatment allocation.

During the screening visit, and after obtaining informed consent, weight, height, waist circumference, blood pressure, and pulse will be measured. Standard blood and urine tests, an oral glucose tolerance test, chest X-ray, and an electrocardiogram will be performed. In addition, volunteers will be interviewed regarding demographic information, medical and family history, dietary habits, and physical activity using questionnaires.

At the run-in visit, participants will retrieve their dairy products and a dietitian will instruct them on how to incorporate 1 daily serving of regular-fat dairy products into their habitual diet. A physical exam will be performed. Participants will be asked to record their food intake for 3 consecutive days (including one weekend day). They will also receive an accelerometer and instructions for use on the same 3-days they record their food intake. Participants will maintain a daily record of consumed dairy products during the run-in periods and throughout the study.

At the baseline and 12-week intervention visits, participants will undergo a hyperinsulinemic-euglycemic clamp to assess systemic insulin sensitivity. In addition, body composition will be measured by dual-energy X-ray absorptiometry and resting energy expenditure by indirect calorimetry.

During the 12-week intervention, participants will be provided with the study products and instructed to consume 2-3 servings/day of regular fat milk, yogurt or cheese. Serving sizes will be 250 mL milk, 175 g yogurt, and 50 g cheese. The dietitian will instruct participants individually on how to incorporate the dairy products into their habitual diets by reducing the intake of other foods of equivalent caloric content and complementary nutrient density to maintain stable body weight. No additional dietary changes will be recommended.

At the monthly follow-up visits, weight, blood pressure, and pulse will be measured. In addition, participants will complete questionnaires about their health and physical activity. At each visit, they will be asked to track their food intake for 3 consecutive days (including one weekend day) using a mobile application on their smartphone or, if not possible, in written food diaries. Additionally, a blood sample will be collected. On the second monthly visit, they will receive an accelerometer and instructions for use on the same 3 days they record their food intake for the 12-week visit.

At the final follow-up visit, participants' weight, blood pressure, and pulse will be measured, and they will complete questionnaires regarding their health and activity. They will also undergo an oral glucose tolerance test and blood tests, as described for the screening visit.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 30 and 65 years,
* Able to provide informed consent,
* Stable weight and dietary habits over a period of 3 months (assessed though questions included in the screening questionnaire regarding changes in weight and dietary habits over the past three months from the date of the screening visit),
* Body mass index of 25-40 kg/m2,
* Waist circumference will follow the International Diabetes Federation ethnic-specific definition (≥94 cm for Europid males, ≥90 cm for Asian males, ≥80 cm for females),
* One or more indicators of prediabetes:

  1. 5.7-6.4% HbA1c
  2. fasting 5.6-6.9 mmol/L glucose, or
  3. 7.8-11.0 mmol/L glucose at 2-hour oral glucose tolerance test (OGTT)

Exclusion Criteria:

* Current smokers,
* Pregnant or planning to become pregnant in the next 6 months,
* Breastfeeding,
* Participation in a weight loss program in the past 3 months,
* Dairy allergy or lactose intolerance,
* Any diagnosed eating disorders,
* Substance abuse (drugs or alcohol >3 drinks/day),
* Diagnosed medical conditions such as cardiovascular disease, anemia, kidney disease, liver disease and any cancer, other than skin, within 5 years.
* Diabetes diagnosis,
* Abnormal electrocardiogram or chest X-Ray,
* Treatment with diuretics, certain β-blockers, bronchodilators, daily nonsteroidal anti-inflammatory drugs, anticoagulants or antiplatelet agents (except prophylactic aspirin 81 mg/d), antianginals, antiarrhythmics, oral steroids, or other medications known to affect glucose metabolism,
* Refusal to temporarily stop taking supplements (minerals, micronutrients, herbal remedies),
* Serum creatinine > 120 µmol/L,
* Hemoglobin < 120 g/L,
* Liver function tests ≥ 3× upper limit,
* Positive viral serology,
* Inaccessible veins.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in whole-body insulin sensitivity | 12 weeks
  Change in whole-body insulin sensitivity as measured by glucose infusion rate during the last 30 min of a hyperinsulinemic-euglycemic clamp divided by serum insulin concentration at the same period (M/I)

SECONDARY OUTCOMES:
Change in glucose tolerance | 13 weeks
  Change in glucose tolerance as measured by plasma glucose concentration at 2-h oral glucose tolerance test
Change in Matsuda index | 13 weeks
  Change in Matsuda index as measured by plasma glucose and insulin concentration during an oral glucose tolerance test
Change in Insulinogenic index | 13 weeks
  Change in Insulinogenic index as measured by the ratio of serum c-peptide concentration and plasma glucose at 30 min minus 0 min during an oral glucose tolerance test
Change in oral disposition index | 13 weeks
  Change in oral disposition index as measured by the product of the Matsuda index and Insulinogenic index
Change in Homeostatic Model Assessment for Insulin Resistance | 13 weeks
  Change in Homeostatic Model Assessment for Insulin Resistance as calculated from fasting glucose and insulin concentration
Change in glycated hemoglobin | 13 weeks
  Change in fasting serum glycated hemoglobin percent
Change in total lean body mass | 12 weeks
  Change in total lean body mass as measured by dual-energy X-ray absorptiometry
Change in total fat mass | 12 weeks
  Change in total fat mass as measured by dual-energy X-ray absorptiometry
Change in visceral fat mass | 12 weeks
  Change in visceral fat mass as estimated by dual-energy X-ray absorptiometry
Change in systolic blood pressure | 12 weeks
  Change in systolic blood pressure as measured by automated blood pressure monitor.
Change in diastolic blood pressure | 12 weeks
  Change in diastolic blood pressure as measured by automated blood pressure monitor.
Change in lipid profile | 12 weeks
  Change in total, LDL-cholesterol as measured as calculated from fasting serum total cholesterol, HDL-cholesterol, and triglycerides

OTHER OUTCOMES:
Change in resting energy expenditure | 12 weeks
  Change in resting energy expenditure as measured by indirect calorimetry
Change in total energy expenditure | 12 weeks
  Change in total energy expenditure as measured by accelerometry
Change in metabolic equivalent of task | 12 weeks
  Change in metabolic equivalent of task as measured by accelerometry
Change in total energy intake | 12 weeks
  Change in total energy intake as calculated from 3-d food records

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Burgos, PhD, Principal Investigator — McGill University
Locations (1):
- RI-MUHC, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No